CLINICAL TRIAL: NCT03890562
Title: Assessing the Effects of Auricular Acupressure on Newborn Behaviors and Withdrawal Signs in Newborns With Neonatal Abstinence Syndrome: A Pilot Study
Brief Title: Assessing the Effects of Auricular Acupressure on Newborns With NAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20006825
Record Dates: First submitted 2018-10-18; First posted 2019-03-26 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: acupressure
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Intervention Model Description: This feasibility study is a single group longitudinal pretest/posttest design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auricular acupressure for NAS infants (Experimental): Auricular acupressure will be applied to five specific acupressure points using a stainless-steel acupressure probe. The five auricular points are: (1) Shen Men, 2) Sympathetic, (3) Kidney, (4) Lung, and (5) Liver. (Tyme, 2001). These sites have been identified by the National Acupuncture Detoxification Association and used for the treatment of withdrawal in adults.
  Interventions: Other: Auricular acupressure

INTERVENTIONS:
Other: Auricular acupressure — Auricular acupressure will be applied to five specific acupressure points using a stainless-steel acupressure probe. The five auricular points are: (1) Shen Men, 2) Sympathetic, (3) Kidney, (4) Lung, and (5) Liver. (Tyme, 2001). These sites have been identified by the National Acupuncture Detoxification Association and used for the treatment of withdrawal in adults.

SUMMARY:
This study will determine the feasibility of using auricular acupressure as an intervention in newborns with neonatal abstinence syndrome(NAS). Auricular acupuncture has been used as an intervention in adults in withdrawal by the National Acupuncture Detoxification Association with good results. The same points on the ear used by National Acupuncture Detoxification Association (NADA) will be used in this intervention using a spring-loaded microprobe to apply minimal pressure instead of needles.

The purpose of this study is to identify barriers to recruiting newborns with NAS; to identify newborn behaviors during the intervention that determine tolerance of the intervention, and to compare results of vitals signs and withdrawal scores prior to intervention and post-intervention.

DETAILED DESCRIPTION:
After Institutional Review Board (IRB) approval, the Primary Investigator (PI) will make daily calls to the units to ascertain whether any newborns have been admitted with a positive drug screen. The researcher will go to the mother's private room after delivery to explain the study. Consents and demographic data will be acquired. The PI will make daily calls to the units to ascertain whether the consented newborns have started on treatment for signs of withdrawal. Before each intervention visit, the PI will call the unit to confirm the newborns feeding schedule with the assigned nurse and arrange for a convenient time to perform the intervention. The intervention will begin on day 1 of pharmacological treatment for withdrawal signs of NAS by the medical staff. The intervention will be provided six times over a 2-week period on day 1,3,5,7,9, and 11 of treatment as recommended by the consulting acupuncturist.

On the day of the intervention the PI will arrive 45 minutes prior to the feeding to perform the following (1) scrub in, (2) set up the secluded area for treatment if infant is not in a private room, (3) transport the newborn to the private/secluded area in the nursery/Neonatal Intensive Care Unit (NICU) if with the mother or in one of the nurseries, (4) perform vital signs (about 3 minutes) and assess ears for any signs of redness or bruising, (5) implement the intervention (approximately 5 minutes), and (6) perform vital signs 5 minutes' post-intervention with post-assessment of ears for any signs of redness or bruising.

Acupressure will be implemented by the PI, using a stainless steel spring-loaded probe to apply small amounts of pressure to the 5 points on the newborn's inner earlobe. The stainless-steel probe will be thoroughly cleaned with alcohol between each newborn. Pressure is given over a 30 second period for each site on the ear and then repeated on the opposite ear. The proposed study will include a fixed intervention as the same intervention will be given to all participants in the treatment group.

The behaviors exhibited by the newborn during intervention will be recorded. Distress signs will be monitored. If they continue for greater than a minute or impede the successful implementation of the intervention, then the intervention will be stopped. The newborn will be soothed and comforted for no greater than ten minutes. If calm after soothing, then intervention will proceed. If the same distress signs are exhibited again, then the intervention will be stopped for the day.

Five minutes' post-intervention the PI will reassess vital signs. The Modified Finnegan Scoring Scale (MFSS) will be taken from the chart for the assessment prior to the intervention and scores immediately post-intervention. Infants who were removed from the mother's room will be returned. Total time for intervention infants should be approximately 35-40 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 36 weeks gestation
* Newborns with positive drug screen and initiation of treatment for withdrawal

Exclusion Criteria:

* Prematurity (< 36 weeks' gestation)
* Any major disease/ illness at birth (e.g. sepsis, necrotizing enterocolitis, gastroenteritis, respiratory disease, cardiac anomalies, anatomical malformation of ears) that could potentially confound the withdrawal symptoms

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited compared to number actually enrolled | Beginning with IRB approval and ending when last eligible newborn completes the intervention. 6 months from IRB approval
  The study will collect data on the difficulty or lack thereof in recruiting the participants for the proposed study. How many mothers of newborns with withdrawal symptoms were approached to participate, agreed to participate, or refused to allow their newborn to be a part of the study? If the mother refused, why did she refuse.

SECONDARY OUTCOMES:
Rate of participant (newborn) study completion | Beginning with first signed consent form and ending when last eligible newborn completes the intervention. about 6 months from first signed consent form
  Number of newborns who completed the final study visit compared to total number of signed consent forms signaling that newborns were enrolled the study

OTHER OUTCOMES:
List of behaviors exhibited by newborns with NAS during auricular acupressure intervention | Beginning with first intervention and ending when last eligible newborn completes the intervention. about 6 months from first intervention
  Newborn behaviors will be recorded during each of the 6 auricular intervention. Behaviors will be logged and noted as indicating distress or indicating tolerance. Behaviors will be compared across all newborns in study.
The Modified Finnegan Score Scale numbers will decrease following intervention. | changes from baseline through day 11
  The Modified Finnegan is a paper and pencil instrument that assesses three major newborn systems: (1) the central nervous system, (2) metabolic/respiratory/vasomotor system, and (3) the gastrointestinal system to quantify withdrawal symptoms with a score of 8 or greater indicating significant withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brown, PhD, RN, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Result] Finnegan LP, Connaughton JF Jr, Kron RE, Emich JP. Neonatal abstinence syndrome: assessment and management. Addict Dis. 1975;2(1-2):141-58. PMID 1163358
- [Result] Tyme, L. (2001). Student Manual on the Fundamentals of Traditional Oriental Medicine (4th edition). Living Earth Enterprises, CA.
- [Result] Warnock F, Sandrin D. Comprehensive description of newborn distress behavior in response to acute pain (newborn male circumcision). Pain. 2004 Feb;107(3):242-255. doi: 10.1016/j.pain.2003.11.006. PMID 14736587